CLINICAL TRIAL: NCT02155023
Title: An Open, Single-centre, Non-controlled Feasibility Study to Determine the Optimal Calibration Method for Glucose Sensors Used for Continuous Glucose Monitoring in Patients With Type 1 Diabetes
Brief Title: Feasibility Study to Determine the Optimal Calibration Method for Glucose Sensors
Acronym: REACT4SENSOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: REACTforSENSOR
Record Dates: First submitted 2014-02-07; First posted 2014-06-04 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine; Insulin Detemir; Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Insulin dosing and glucose sensors (Experimental): To test the glucose sensors different levels of glycemia are needed. To provoke different glycemic levels the following intervention will be performed: Lunch (with fast glucose absorption characteristics) will be served. Up to 30 minutes after the usual insulin dosing time, the subjects will take his/her lunch dose of insulin adjusted to the chosen lunch plus additional approximately 25% (in the range of 0-50% according to the discretion of the Investigator) of insulin - in order to provoke moderate postprandial hypoglycaemia with glucose values < 70 mg/dl.
  Interventions: Drug: Insulin dosing; Device: Glucose sensors IR-Glucose Reader (Joanneum Research, Austria), IR-CGM (IMM, Germany)

INTERVENTIONS:
Drug: Insulin dosing
  Other Names: Subjects will use their daily usual insulin:; Lantus; Levemir; Humalog; Novorapid; Sensors:; IR-Glucose Reader (Joanneum Research, Austria); IR-CGM (IMM, Germany)
Device: Glucose sensors IR-Glucose Reader (Joanneum Research, Austria), IR-CGM (IMM, Germany)

SUMMARY:
Two new glucose sensors (IR-Glucose Reader (Joanneum Research, Austria), IR-CGM (IMM, Germany)) will be investigated to determine the optimal calibration method in patients with type 1 diabetes

DETAILED DESCRIPTION:
The subjects (Type 1 diabetes) will stay at the Clinical Research Centre for the whole period of the investigation (12 hours).

Continuous blood glucose monitoring will be performed using the IR-Glucose Reader system and/or the IR-CGM system based on microdialysis. In parallel blood glucose measurements will be performed every 15 min as reference. The measurements of the sensors will be calibrated with different schemes and the difference between the calibrated glucose readings and the reference blood glucose values will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained after being advised of the nature of the study
* Male or female aged 18 to 75 years (both inclusive)
* The subject has Type 1 diabetes (as defined by WHO) for at least 24 months
* Body Mass Index (BMI) <= 35 kg/m2

Exclusion Criteria:

* Subject is actively enrolled in another clinical trial or took part in a study within 30 days
* Experienced recurrent severe hypoglycaemic unawareness (as judged by the investigator)
* A history of drug or alcohol dependence
* Positive result for HIV antibodies
* Positive result for Hepatitis B antigen or Hepatitis C antibodies
* Any other significant concomitant disease such as endocrine, cardiac, neurological, malignant, other pancreatic disease or uncontrolled hypertension as judged by the investigator
* Patient is pregnant, or breast feeding during the period of the study
* Patient donated blood in the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
difference between calibrated measurements and reference | 12 hours
  The calibrated sensor signals will be compared with the reference blood glucose values. The difference between the calibrated sensor signal and the reference values will be calculated (which corresponds to the error of the sensor signal)

SECONDARY OUTCOMES:
evaluate necessary run-in procedures by assessment of error over time | 12 hours
  Once the difference between sensor signal and the reference values is calculated these values will be investigated by looking at the data over time which enables to detect a possible change of the difference.

OTHER OUTCOMES:
Distribution of the glucose values | 12 hours
  The glucose sensors will be tested over a range of different reference glucose values. The distribution of the glucose values (hypo-normo-hyperglycaemia) will be taken into account when calculating the difference (error) between the sensor- and reference value.
Malfunction of the systems | 12 hours
  Based on the fact that the sensors are in a very early development stage possible malfunctions of the sensor systems will be recorded and categorized to: mechanical, electrical, software and other malfunctions

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Pieber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

REFERENCES:
- See also: Website of the project which is funded by the European Commission — http://www.reaction-project.eu